CLINICAL TRIAL: NCT04211259
Title: The Prophylactic Use of Loratadine for Granulocyte-Colony Stimulating Factor (G-CSF) Induced Bone Pain in Multiple Myeloma Patients Undergoing Stem Cell Mobilization
Brief Title: Loratadine for the Reduction of G-CSF Induced Bone Pain in Patients With Multiple Myeloma Undergoing Stem Cell Mobilization
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mansi Shah, MD, Assistant Professor of Medicine, Rutgers Cancer Institute of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 011910; NCI-2019-07795 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2019001846; Pro2019001846 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (loratadine) (Experimental): Beginning 5 days before the first dose of standard of care filgrastim, patients receive loratadine PO QD. Treatment continues until 5 days after completion of stem cell mobilization in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Loratadine; Other: Questionnaire Administration
- Cohort II (placebo) (Placebo Comparator): Beginning 5 days before the first dose of standard of care filgrastim, patients receive placebo PO QD. Treatment continues until 5 days after completion of stem cell mobilization in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Loratadine — Given PO
  Other Names: Claritin
  Arms: Cohort I (loratadine)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Cohort II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial studies how well loratadine works in reducing granulocyte-colony stimulating factor (G-CSF) induced bone pain in patients with multiple myeloma who are undergoing stem cell mobilization. Loratadine is an antihistamine that may help to reduce or control bone pain during the process of stem cell collection in patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of the second-generation antihistamine, loratadine, as prophylaxis for filgrastim (i.e., Neupogen, Zarxio) induced bone pain during stem cell mobilization in multiple myeloma patients.

SECONDARY OBJECTIVES:

I. To examine the frequency and quantity of supportive analgesic medications needed in addition to loratadine or placebo for filgrastim induced bone pain.

II. To identify risk factors associated with developing filgrastim induced bone pain.

OUTLINE: Patients are randomized to 1 of 2 cohorts.

COHORT I: Beginning 5 days before the first dose of standard of care filgrastim, patients receive loratadine orally (PO) once daily (QD). Treatment continues until 5 days after completion of stem cell mobilization in the absence of disease progression or unacceptable toxicity.

COHORT II: Beginning 5 days before the first dose of standard of care filgrastim, patients receive placebo PO QD. Treatment continues until 5 days after completion of stem cell mobilization in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able to provide informed consent
* Patients with confirmed diagnosis of multiple myeloma
* Able to swallow and retain oral medication
* All ethnic groups are eligible

Exclusion Criteria:

* Non-English speaking person
* Patients undergoing haploidentical allogeneic hematopoietic stem cell transplant
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds
* Any medical complications or conditions that would, in the investigator's judgement, interfere with full participation in the study
* On therapeutic dose of aspirin (doses greater than 81 mg) within 7 days prior to the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean pain level for each group following therapy | Baseline up to 5 days after completion of stem cell mobilization
  Pain severity will be measured at baseline and following treatment using a 10-point scale, with higher numbers indicating greater degrees of pain. Will compare the difference in mean pain level for each group following therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mansi R. Shah, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No